CLINICAL TRIAL: NCT07198347
Title: A Randomized, Double-blind, Active-controlled, Parallel-group, Multicenter, Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of AG2001 in Patients With Acute Bronchitis
Brief Title: Efficacy and Safety of AG2001 in Patients With Acute Bronchitis
Acronym: AG2001 P3
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ahn-Gook Pharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AG2001 P3; AG2001 P3 (Other: Ahngook Pharm)
Record Dates: First submitted 2025-09-15; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Acute Bronchitis
Keywords: acute bronchitis; Cough; Sputum
MeSH Terms: conditions — Bronchitis; Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AG2001 (Experimental): Participants receive AG2001 with matching placebos, administered orally three times daily for 7 days.
  Interventions: Drug: AG2001
- AG20011 (Active Comparator): Participants receive AG20011 with matching placebos, administered orally three times daily for 7 days.
  Interventions: Drug: AG20011
- AG20012 (Active Comparator): Participants receive AG20012 with matching placebos, administered orally three times daily for 7 days.
  Interventions: Drug: AG20012

INTERVENTIONS:
Drug: AG2001 — Oral administration, three times daily for 7 days.
  Arms: AG2001
Drug: AG20011 — Oral administration, three times daily for 7 days.
  Arms: AG20011
Drug: AG20012 — Oral administration, three times daily for 7 days.
  Arms: AG20012

SUMMARY:
This is a Phase 3, randomized, double-blind, active-controlled clinical trial designed to evaluate the efficacy and safety of AG2001 in patients with acute bronchitis. The primary objective is to demonstrate the superiority of AG2001 over two active comparators based on the change in Bronchitis Severity Score (BSS) at Day 4.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥19 years to <65 years old
2. Subjects who present symptoms of Acute Bronchitis with cough and sputum symptoms within 48 hours prior the randomization visit(Visit 2) who satisfy the following

   * Total Bronchitis Severity Scale ≥ 5
   * Total Bronchitis Severity Scale sputum score ≥ 2
3. Subjects who without fever(condensed body temperature standard: less than 38.5°C) prior to randomization visit(Visit 2)
4. Subjects who present symptoms of Acute Bronchitis with cough less then 2 weeks prior to randomization visit(Visit 2)
5. Written consent voluntarily to participate who can understand the information provided in this clinical trial

Exclusion Criteria:

* Chronic respiratory diseases (e.g., COPD, asthma, pneumonia, tuberculosis, lung cancer)
* Clinically significant hepatic, renal, cardiovascular, or neurological disorders
* Use of prohibited medications (e.g., antibiotics, antivirals, corticosteroids) within the washout period
* Positive test for hepatitis B, hepatitis C, or HIV
* Pregnant or breastfeeding women
* Any condition deemed inappropriate by the investigator

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Bronchitis Severity Score (BSS) from Baseline to Day 4 | Baseline to Day 4
  The difference in BSS total score compared between treatment and comparator groups.

SECONDARY OUTCOMES:
Change in Bronchitis Severity Score (BSS) from Baseline to Day 7 | Baseline to Day 7
  Evaluation of the change in BSS total score between baseline and Day 7.
Change in BSS Subscale Scores (cough, sputum, etc.) at Day 4 and Day 7 | Baseline to Day 4 and Day 7
  Assessment of individual BSS subscale scores including cough and sputum severity.
Proportion of BSS Responders at Day 4 and Day 7 | Baseline to Day 4 and Day 7
  Percentage of participants achieving predefined responder criteria based on BSS score improvement.
Change in Integrative Medicine Outcome Scale (IMOS) | Baseline to Day 4 and Day 7
  Evaluation of IMOS scores as secondary endpoints.
Change in Integrative Medicine Patient Satisfaction Scale (IMPSS) | Baseline to Day 4 and Day 7
  Evaluation of IMPSS scores as secondary endpoints.
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 30 days after last dose
  Safety evaluation including the number and proportion of participants experiencing AEs and SAEs.

IPD SHARING:
Plan to Share IPD: No